CLINICAL TRIAL: NCT01909102
Title: The ACTonHEART Study: a Randomized Controlled Clinical Trial of Acceptance and Commitment Therapy in Cardiac Patients
Brief Title: The ACTonHEART Study: Design of a Randomized Controlled Clinical Trial of Acceptance and Commitment Therapy for Cardiac Patients
Acronym: ACTonHEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03C301
Record Dates: First submitted 2013-07-17; First posted 2013-07-26 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Cardiovascular Diseases
Keywords: Acceptance and Commitment Therapy; Cardiac rehabilitation
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT-based intervention (Experimental): The ACT-based intervention integrates educational topics on heart healthy behaviours with mindfulness and acceptance training regarding difficult thoughts and feelings, clarification of health-related values and commitment to behave in the valued direction while contacting difficult experiences.
  Interventions: Behavioral: ACT-based intervention; Behavioral: usual care
- Usual care (Active Comparator): Usual care is based on current guidelines for the long-term multi-disciplinary rehabilitation and prevention of cardiac patients.
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: ACT-based intervention
  Arms: ACT-based intervention
Behavioral: usual care

SUMMARY:
The study will determine whether a brief intervention program based on Acceptance and Commitment Therapy can be effective for the reduction of modifiable risk factors and improvement of psychological well-being in patients referred to cardiac rehabilitation

DETAILED DESCRIPTION:
The Acceptance and Commitment Therapy is a mindfulness-based intervention which efficacy has been proven in the treatment of depression and anxiety, in stress reduction and in the modification of health- related behaviors in patients with several physical conditions. The application of an acceptance-based program in cardiac patients has revealed high treatment satisfaction and initial evidences of effectiveness in increasing heart-healthy behaviour.

The purpose of the trial is to evaluate the efficacy of a brief group-administered program based on Acceptance and Commitment Therapy in improving patients' ability to address modifiable multiple cardiovascular risk factors and overall psychological well-being, compared with the usual care.

ELIGIBILITY:
Inclusion Criteria:

* having a current diagnosis of ischemic heart disease (IHD)
* being affected by major modifiable cardiovascular risk factors that will be assessed through the INTERHEART Modifiable Risk Score.

Only subjects with a full score >9 will be included in the study.

* between the ages of 18 and 70 years
* fluency in spoken and written Italian language
* expression of written informed consent.

Exclusion Criteria:

* cognitive impairment
* severe psychiatric disorders according to Diagnostic and Statistical Manual-IV TR criteria (APA, 2000).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-08; Primary Completion 2022-03 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Low-density lipoprotein (LDL)cholesterol | Baseline and 12 months
  Change from baseline LDL cholesterol level
Blood pressure | baseline and 12 months
  Change from baseline resting blood pressure (the mean of 2 measures taken 2 minutes apart with a manual sphygmomanometer)
Body Mass Index | baseline and 12 months
  Change from baseline Body Mass Index. It is calculated as weight in kilograms divided by height in meters squared
Psychological Well-Being | Baseline and 12 months
  Change from baseline Psychological Well-Being. It will be measured by the Psychological General Well-Being Inventory. The PGWBI is a self-administered questionnaire composed by six sub-scales: anxiety, depression, positive well-being, self-control, general health and vitality. Higher scores indicate better health.

SECONDARY OUTCOMES:
Health-related quality of life | Baseline and 12 months
  Change from baseline Health-related quality of life. The Short Form-36 questionnaire for evaluation of Quality Of Life is widely used and gives valuable information on Quality Of Life related to health. The patients' Quality Of Life will be assessed through the following eight fractions: physical function, physical role, general health, social function, experience of pain, mental health, emotional role and vitality.
Dietary habits | Baseline and 12 months
  Change from baseline dietary habits. They will be assessed through the Mediterranean diet score, a large-scale diet score based on the inherent characteristics of Mediterranean dietary pattern. Questions focused on the frequency of usual consumption of 11 main components of the Mediterranean diet (nonrefined cereals, fruits, vegetables, potatoes, legumes, olive oil, fish, red meat, poultry, full fat dairy products and alcohol).
Physical activity | Baseline anf 12 months
  Change from baseline physical activity. It will be measured by The International Physical Activity Questionnaire (IPAQ), a self-report questionnaire that assesses the number of days per week and the number of times per day an individual spends doing specific activities.
Smoking cessation | At 1-year follow-up
  Self-report of smoking status
Adherence to medication | Baseline and 12 months
  Change from baseline adherence to medication. The Modified Morisky Scale will be used. It is a eight-item self-reported measure of medication taking.
Exercise capability | Baseline and 12 months
  Change from baseline exercise capability. The exercise capability will be considered as the maximal power (in Watts) reached during an incremental bicycle stress test.

OTHER OUTCOMES:
Psychological inflexibility | Baseline and 12 months
  Change from baseline psychological inflexibility. It will be measured through the Acceptance and Action Questionnaire-II, a self-report 10-item scale.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Castelnuovo, PhD, PsyD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- San Luca Hospital, Istituto Auxologico Italiano, Milan, Italy

REFERENCES:
- [Background] Goodwin CL, Forman EM, Herbert JD, Butryn ML, Ledley GS. A pilot study examining the initial effectiveness of a brief acceptance-based behavior therapy for modifying diet and physical activity among cardiac patients. Behav Modif. 2012 Mar;36(2):199-217. doi: 10.1177/0145445511427770. Epub 2011 Nov 30. PMID 22133992
- [Derived] Spatola CAM, Rapelli G, Giusti EM, Cattivelli R, Goodwin CL, Pietrabissa G, Malfatto G, Facchini M, Cappella EAM, Varallo G, Martino G, Castelnuovo G. Effects of a brief intervention based on Acceptance and Commitment Therapy versus usual care for cardiac rehabilitation patients with coronary heart disease (ACTonHEART): a randomised controlled trial. BMJ Open. 2024 Jun 12;14(6):e084070. doi: 10.1136/bmjopen-2024-084070. PMID 38866567
- [Derived] Spatola CA, Manzoni GM, Castelnuovo G, Malfatto G, Facchini M, Goodwin CL, Baruffi M, Molinari E. The ACTonHEART study: rationale and design of a randomized controlled clinical trial comparing a brief intervention based on Acceptance and Commitment Therapy to usual secondary prevention care of coronary heart disease. Health Qual Life Outcomes. 2014 Feb 19;12:22. doi: 10.1186/1477-7525-12-22. PMID 24552555